CLINICAL TRIAL: NCT07228793
Title: Natural History Prospective Open Clinical and Genetic Study of Patients With EYS-Associated Retinitis Pigmentosa
Brief Title: Natural History Study of Patients With EYS-Associated RP
Acronym: RUS_EYS
Status: Recruiting | Type: Observational
Sponsor: Sensor Technology for Deafblind (Industry)
Collaborators: Russian RetinaFond (Unknown)
Responsible Party: Principal Investigator, Marianna E. Weener, MD, PhD, Medical Center Oftalmika
Other Study IDs: EYS_RUS_2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Retinitis Pigmentosa; Eye Diseases
Keywords: EYS mutation; RP; Retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — peripheral venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vision Cohort 1: Participants with the better eye Screening Visit decimal visual acuity of 0.4 or more and visual field diameter 10 degrees or more in every meridian of the central field.
  Interventions: Diagnostic Test: Whole exome/genome sequencing
- Vision Cohort 2: Participants with the better eye Screening Visit decimal visual acuity 0.15 - 0.35 and visual field diameter less than 10 degrees in any meridian of the central field)
  Interventions: Diagnostic Test: Whole exome/genome sequencing
- Vision Cohort 3: Participants with the better eye Screening Visit decimal visual acuity 0.14 or less.
  Interventions: Diagnostic Test: Whole exome/genome sequencing

INTERVENTIONS:
Diagnostic Test: Whole exome/genome sequencing — Next generation sequencing and segregation analysis or long read sequencing for confirmation of biallelic mutations (in trans-position)

SUMMARY:
This natural history study of patients with EYS mutations from Russia and former CIS (Commonwealth of Independent States) territories will accelerate the development of outcome measures for clinical trials. Sensitive, reliable outcome measures of retinal degeneration will greatly facilitate development of treatments for retinitis pigmentosa due to EYS mutations. This approach helps to develop experimental treatment protocol, and assessing its effectiveness.

The goals and expected impact of this natural history study are to:

1. Describe the natural history of retinal degeneration in patients with biallelic mutations in EYS gene in Russia and former CIS territories.
2. Identify sensitive structural and functional outcome measures to use for future multicenter clinical trials in EYS-related retinal degeneration in Russia and former CIS territories.
3. Identify well-defined subpopulations for future clinical trials of investigative treatments for EYS-related retinal degeneration in Russia and former CIS territories.

DETAILED DESCRIPTION:
1. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the EYS gene over 4 years, as measured using functional, structural, and patient-reported outcome measures
2. Investigate whether structural outcome measures can be validated as surrogates for functional outcomes in individuals with biallelic pathogenic mutations in the EYS gene
3. Evaluate risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with biallelic pathogenic mutations in the EYS gene
4. Evaluate variability and symmetry of left and right eye outcomes over 4 years in individuals with biallelic pathogenic mutations in the EYS gene

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and able to communicate consent during the consent process
2. Ability to return for all study visits over 48 months
3. Age ≥ 18 years
4. Must meet one of the Genetic Screening Criteria, defined below:

Screening Group A: At least 2 disease-causing variants in the EYS gene which are homozygous or heterozygous in trans, based on a report from a clinically-certified lab (or a report from a research lab that has been pre-approved by the Study Committee) Screening Group B: Only 1 disease-causing variant in the EYS gene, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Study Committee) Screening Group C: At least 2 disease-causing variants in the EYS gene which are unknown phase, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Study Committee) Note pertaining to all Screening Groups: if a participant has a variant(s) of unknown significance, he/she would still qualify as long as there is at least 1 disease-causing variant(s) on the EYS gene.

Ocular Inclusion Criteria:

Both eyes must meet all of the following:

1. Clinical diagnosis of retinal dystrophy
2. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging

Exclusion Criteria:

1. Mutations in genes that cause autosomal dominant retinitis pigmentosa (ADRP), X-linked retinitis pigmentosa (RP), or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than EYS.
2. Expected to enter experimental treatment trial at any time during this study
3. History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine)

Ocular exclusion Criteria:

If either eye has any of the following, the participant is not eligible:

* Current vitreous hemorrhage
* Current or any history of rhegmatogenous retinal detachment
* Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia
* History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months
* Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucomatous visual functions changes or nerve changes, or history of glaucoma filtering surgery)
* Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy
* History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function
* History or evidence of active treatment for retinitis pigmentosa that could affect the progression of retinal degeneration, including:
* Any use of ocular stem cell or gene therapy
* Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Screening Visit date)
* Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Screening Visit date is at least 5 times the half-life of the given product)

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential eligibility may be assessed as part of a routine care examination by an investigator prior to obtaining informed consent, as part of usual care, by referral from another physician, or self-referral.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Field Sensitivity | Baseline and every year until study completion (4 years)
  Measured by static perimetry with topographic analysis and assessed by a certified reading center for cohorts 1 and 2.
Change in Retinal Function | Baseline and 4 year follow-up visit.
  Measured by full-field electroretinogram (ERG) amplitudes and timing in response to rod- and cone-specific stimuli for cohorts 1 and 2.

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity | Screening visit and every year until study completion (4 years) for cohort 1&2. Screening visit and 48 month follow-up for cohort 3.
  Measured on Golovina-Sivtsev charts
Change in Mean Retinal Sensitivity | Baseline and every year until study completion (4 years)
  Measured by fundus-guided microperimetry (MP) and assessed by a certified reading center for cohorts 1 and 2.
Change in Best Corrected Low Luminance visual acuity | Screening visit and every year until study completion (4 years) for cohort 1&2. Screening visit and 48 month follow-up for cohort 3.
  Measured by letter score
Change in Contrast Sensitivity Function | Baseline and every year until study completion (4 years).
  Measured by Zebra software for cohorts 1 and 2.
Change in Ellipsoid zone (EZ) area | Baseline and every year until study completion (4 years) for cohorts 1 and 2. Baseline and 4 year follow-up for cohort 3.
  Measured by spectral domain optical coherence tomography (SD-OCT) and assessed by a certified expert
Explore qualitative and quantitative categorization of Fundus Autofluorescence (FAF) pattern | Baseline and every year until study completion (4 years) for cohorts 1 and 2. Baseline and 4 year follow-up for cohort 3.
  Assessed by a certified expert

OTHER OUTCOMES:
Patient Reported Outcomes for Vision Cohorts 1, 2 and 3 | Baseline and 4 year follow-up visit
  Measured by modified MRDQ (Michigan Retinal Degeneration Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Weener, MD, PhD, Principal Investigator — Oftalmic
Locations (1):
- Oftalmic Clinical Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
A de-identified database will be placed in the public domain on the Oftalmic public website after the completion of each protocol and publication of the manuscript.
Supporting Information: CSR
Time Frame: After manuscript is published
Access Criteria: Users accessing data must enter an email address